CLINICAL TRIAL: NCT05493826
Title: Real-world Evidence Study on the Early Use of Cemiplimab in the UK: REACT-CEMI (Real World Evidence of Advanced CSCC Treatment - With CEMIplimab)
Brief Title: Real World Study on the Use of Cemiplimab in Adult Patients in UK
Acronym: REACT-CEMI
Status: Completed | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: DUT0052
Record Dates: First submitted 2022-08-07; First posted 2022-08-09 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Cutaneous Squamous Cell Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Patients treated with cemiplimab for laCSCC or mCSCC who were not suitable for curative surgery or curative radiation
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Non-interventional study based on secondary use of hospital medical record

SUMMARY:
The primary objective is to describe the real-world clinical effectiveness of cemiplimab in patients with locally advanced cutaneous squamous cell carcinoma (laCSCC) or metastatic cutaneous squamous cell carcinoma (mCSCC) treated in routine clinical practice.

DETAILED DESCRIPTION:
Patients initiating treatment with cemiplimab in the UK between 2nd July 2019 and 30th November 2020, will be followed for a minimum of 12 and a maximum of 36 months from initiation of cemiplimab.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >=18 years at initiation of cemiplimab.
* Patients treated with >=1 dose of cemiplimab for laCSCC or mCSCC who were not suitable for curative surgery or curative radiation according to routine practice.
* Patients initiating treatment with cemiplimab in the UK between 2nd July 2019 and 30th November 2020.

Exclusion Criteria:

* Patients who are known to have opted out of participation in any research (as required for compliance with GDPR).
* Patients participating in any form of investigative study (e.g., clinical trials) during the post-index observation period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with cemiplimab for laCSCC or mCSCC who were not suitable for curative surgery or curative radiation
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) within 12 months post initiation of cemiplimab | 12 months
  ORR, defined as the proportion of patients who have a partial or complete response to cemiplimab based on an assessment according to routine practice, as documented in medical records

SECONDARY OUTCOMES:
ORR within 6 months post initiation of cemiplimab | 6 months
Real-world best response within 6- and 12-months post initiation of cemiplimab | 6 months, 12 months
  Real-world best response, defined as the best response to cemiplimab observed during the observation period.
Time to best response | From initiation of cemiplimab until data collection or death, whichever is earliest, up to 36 months
  The best response to cemiplimab observed during the observation period
Time to partial response | From initiation of cemiplimab until data collection or death, whichever is earliest, up to 36 months
  Time to partial response, defined as time from cemiplimab initiation until the first documentation of a partial response based on assessment according to routine practice, as documented in medical records.
Time to complete response | From initiation of cemiplimab until data collection or death, whichever is earliest, up to 36 months
  Time to complete response, defined as time from cemiplimab initiation until the first documentation of a complete response based on assessment according to routine practice, as documented in medical records.
Disease control rate (DCR) within 6 and 12 months post initiation of cemiplimab | 6 months, 12 months
  DCR, defined as the proportion of patients who have a complete response, partial response or stable disease based on an assessment according to routine practice, as documented in medical records
Duration of response (DoR) | From initiation of cemiplimab until data collection or death, whichever is earliest, up to 36 months
  DoR, defined as the time from the first documentation of a complete or partial response to cemiplimab in medical records until first documentation of disease progression or death
Duration of treatment (DoT) | From initiation of cemiplimab until data collection or death, whichever is earliest, up to 36 months
  DoT, defined as the time from cemiplimab initiation to the documented date of treatment discontinuation.
Real-world progression-free survival (rwPFS) | From initiation of cemiplimab until data collection or death, whichever is earliest, up to 36 months
  rwPFS, defined as the time from cemiplimab initiation to date of disease progression or death as recorded in the medical records
Overall survival (OS) | From initiation of cemiplimab until data collection or death, whichever is earliest, up to 36 months
  OS, defined as the time from cemiplimab initiation to date of death from any cause.
Demographics | Baseline
  Age, Sex, Ethnicity
Medical history | Baseline
  Co-morbidities, Eastern Cooperative Oncology Group performance status, Stage of disease, Primary CSCC lesion disease site and date diagnosed (where available), Time from diagnosis of primary disease to diagnosis of laCSCC or mCSCC not suitable for curative surgery or curative radiotherapy (where available)
Previous treatments | Baseline
  Previous treatments for cemiplimab index CSCC lesion(s) during the pre-index observation period, Previous treatments for cemiplimab non-index CSCC lesion(s) during the pre-index observation period, Previous treatments for any prior skin malignancies during the pre-index observation period
Clinical characteristics outcome | Baseline
  Proportion of patients treated with antibiotics in the 6 wks prior to or 6 wks post-initiation of cemiplimab, Proportion of patients with immunocompromised status and treatment history incl. any concomitant therapy, Proportion of patients with a history of organ transplantation, Frequency and distribution of prior organ transplantations by type, Frequency and distribution of prior malignancies overall and by type, Type of Multidisciplinary team review and referral prior to laCSCC/mCSCC diagnosis
Number of cemiplimab infusions | From initiation of cemiplimab until data collection or death, whichever is earliest, up to 36 months
Proportion of patients where cemiplimab treatment was interrupted, overall and by reason for interruption | From initiation of cemiplimab until data collection or death, whichever is earliest, up to 36 months
Proportion of patients permanently discontinuing treatment, overall and by reason for discontinuation | From initiation of cemiplimab until data collection or death, whichever is earliest, up to 36 months
Distribution of cemiplimab dose administered at initiation | From initiation of cemiplimab until data collection or death, whichever is earliest, up to 36 months
Proportion of patients experiencing immune-related adverse reactions (irARs) of any grade (where reported in notes) | From initiation of cemiplimab until data collection or death, whichever is earliest, up to 36 months
  irAR, defined as treatment-related, immune-related adverse events (as defined by local investigator)
Proportion of patients with cemiplimab treatment interruptions due to experiencing irARs | From initiation of cemiplimab until data collection or death, whichever is earliest, up to 36 months
Duration of treatment interruption for patients experiencing irARs | From initiation of cemiplimab until data collection or death, whichever is earliest, up to 36 months
Proportion of patients treated with anti-inflammatory drugs (e.g., steroids) for irARs, overall and by type of irAR | From initiation of cemiplimab until data collection or death, whichever is earliest, up to 36 months
Initial dose of anti-inflammatory drug (e.g., steroids) used to treat irARs at onset of irARs and for the duration of irARs by steroid type | From initiation of cemiplimab until data collection or death, whichever is earliest, up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences and Operations, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis UK, Reading, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org